CLINICAL TRIAL: NCT02657564
Title: The Renal Safety of Bowel Preparation With Polyethylene Glycol for Colonoscopy: A Prospective Cohort Study
Brief Title: Renal Safety of Bowel Preparation With Polyethylene Glycol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evergreen General Hospital, Taiwan (Other)
Responsible Party: Principal Investigator, Chi-Liang Cheng, Assistant Professor, Evergreen General Hospital, Taiwan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ZEH-2016-1
Record Dates: First submitted 2015-11-17; First posted 2016-01-18 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Polyethylene Glycols; klean prep

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Polyethylene glycol (PEG) (Other): 3-L polyethylene glycol (PEG) is provided for colonoscopy preparation. Patients receive blood tests for renal function and electrolytes before and after colonoscopy.
  Interventions: Drug: Polyethylene glycol (PEG)

INTERVENTIONS:
Drug: Polyethylene glycol (PEG) — Participants receive blood tests for serum creatinine and electrolytes (Ca, P, Cl, Mg, Na, K) before and after taking polythylene glycol.
  Other Names: Klean-Prep

SUMMARY:
This study evaluates the changes of renal function after taking bowel cleansing agent polyethylene glycol for elective colonoscopy.

DETAILED DESCRIPTION:
Polyethylene glycol (PEG) is the most commonly used bowel cleansing agent for colonoscopy in the world.

PEGs are non-absorbable isosmotic solutions that pass through the bowel without net absorption or secretion. Significant fluid and electrolyte shifts are therefore attenuated.

However, several studies have shown that PEG may also impair renal function. One recent population-based study reported that the use of PEG was associated with an increased risk of acute kidney injury.

The renal safety of PEG in Taiwanese patient has not been reported.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 40 yrs of age or older scheduled for elective colonoscopy.

Exclusion Criteria:

* Severely reduced kidney function (eGFR] <30 mL/min/1.73 m2)
* Serum electrolyte abnormalities at screening
* Uncontrolled congestive heart failure (American Heart Association Classification III or IV)
* Unstable angina
* Untreated dysrhythmia
* Myocardial infarction, percutaneous transluminal coronary angioplasty, or coronary artery bypass graft surgery within the previous 3 months
* Ascites
* Current acute exacerbation of chronic inflammatory bowel disease
* Toxic colitis or toxic megacolon
* Ileus and/or acute obstruction or perforation
* Ileostomy
* Right or transverse colostomy
* Subtotal colectomy with ileosigmoidostomy

  * 50% of colon removed
* Idiopathic pseudo-obstruction
* History of gastric stapling or bypass procedure
* Difficulties swallowing
* Treatment with an investigational drug or product
* Participation in a drug study within 30 days prior to receiving study medication
* Treatment with another bowel preparation within 21 days prior to colonoscopy
* Known allergy or hypersensitivity to PEG solution

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1237 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chiliang Cheng, MD, Principal Investigator — Zhongli Evergreen General Hospital, Taiwan
Locations (1):
- Evergreen General Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Polyethylene Glycol (PEG)
Started | 1237
Completed | 1163
Not Completed | 74

BASELINE CHARACTERISTICS:
Groups:
- Polyethylene Glycol (PEG): 3L polyethylene glycol (PEG) is provided for colonoscopy preparation. Patients receive blood tests for renal function and electrolytes before and after colonoscopy.
  3L Polyethylene glycol (PEG): Participants receive blood tests for serum creatinine and electrolytes (Ca, P, Cl, Mg, Na, K) before and after taking polythylene glycol.
Arm/Group | Polyethylene Glycol (PEG)
Number analyzed (Participants) | 1163
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 623
  Male | 540
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Renal Injury Which Included Acute Renal Dysfunction and Acute Kidney Injury
Description: The screening visit (visit 1) induced a blood specimen for serum chemistry analysis. Immediately before the colonoscopy, study staff collected blood specimens for chemistry analysis (visit 2). The patients returned within 28 days after the colonoscopy for a final renal test (visit 3). Patients with a ≥30% increase above baseline creatinine levels during visit 2 or 3 were followed every 2-4 weeks until a peak level was detected (visit 4 and beyond).The serum creatinine level on visit 1 was recorded as the baseline renal function. The presence of renal injuries was determined by the highest serum creatinine level noted during the study period and included acute renal dysfunction, defined as a 30-49% increase above the baseline creatinine level, and acute kidney injury, defined as a ≥50% increase above the baseline serum creatinine. Number of participants with acute renal injury which included acute renal dysfunction and acute kidney injury will be recorded.
Time Frame: The durations between visits 1-2 and visits 2-3 were within 28 days, respectively. Patients with a ≥30% increase above the baseline serum creatinine levels during visit 2 or 3 were followed every 2-4 weeks until a peak level of creatinine was detected.
Measure: Number; unit: participants
Groups:
- Polyethylene Glycol (PEG): A total of 1,163 patients completed the study protocol in which 3-L polyethylene glycol was used as colonoscopy preparation.
Arm/Group | Polyethylene Glycol (PEG)
Number analyzed (Participants) | 1163
participants | 32

2. Secondary Outcome: Number of Participants With Acute Electrolyte Disturbance (Including Serum Caclium, Phosphate, Sodium, Potassium, Chloride, and Magnesium).
Description: The screening visit (visit 1) induced a blood specimen for serum chemistry analysis. Immediately before the colonoscopy, study staff collected blood specimens for chemistry analysis (visit 2). The patients returned within 28 days after the colonoscopy for a final renal safety evaluation (visit 3). Patients with electrolyte abnormalities during visit 2 or visit 3 were followed every 2-4 weeks until serum electrolyte values returned to normal.
Time Frame: The durations between visits 1-2 and visits 2-3 were within 28 days, respectively. Patients with electrolyte abnormalities during visit 2 or visit 3 were followed every 2-4 weeks until serum electrolyte values returned to normal.
Measure: Count of Participants; unit: Participants
Arm/Group | Polyethylene Glycol (PEG)
Number analyzed (Participants) | 1163
Participants | 447

ADVERSE EVENTS:
Time Frame: Colonoscopy related complication was observed during and within one month after colonoscopy. Patient with acute renal injury were followed every 2-4 weeks until a peak level of creatinine was detected.Renal recovery was examined every month after the peak creatinine level was reached. Patients with electrolyte abnormalities during visit 2 or visit 3 were followed every 2-4 weeks until serum electrolyte values returned to normal.
Arm/Group | Polyethylene Glycol (PEG)
All-Cause Mortality (participants affected / at risk) | 0/1163
Serious Adverse Events (participants affected / at risk) | 0/1163
Other Adverse Events (participants affected / at risk) | 350/1163
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Polyethylene Glycol (PEG) (N=1163)
Any Electrolyte Abnormality (General disorders) | 350 (350) — Acute electrolyte abnormalities included hypocalcemia, hypophosphatemia, and hyperchloremia.
Hypocalcemia (General disorders) | 300 (300)
Hypophosphatemia (General disorders) | 139 (139)
Hyperchloremia (General disorders) | 77 (77)
Hypokalemia (General disorders) | 52 (52)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-11-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT02657564/Prot_000.pdf
  • Statistical Analysis Plan (2015-11-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT02657564/SAP_001.pdf